CLINICAL TRIAL: NCT05019014
Title: Olfactory Deficits in Neurologic Disease
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark William Albers, Frank Wilkens and Family Endowed Scholar/ Asst. Prof. Neurology, Massachusetts General Hospital
Other Study IDs: 2011P001296
Record Dates: First submitted 2017-04-07; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease; Traumatic Brain Injury; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Lewy Body Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Brain Injuries, Traumatic; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Lewy Body Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurodegenerative disease: Participants with a diagnosis of Probable Alzheimer's Disease, prodromal Alzheimer's Disease, Frontotemporal Dementia, Mild Cognitive Impairment, Dementia with Lewy Bodies, mild and moderate/severe TBI, and familial or sporadic ALS per El Escorial Criteria or individuals with known gene mutations associated with ALS.
- Age-matched controls: Healthy participants with no diagnosis.

SUMMARY:
The goal of this study is to examine olfactory function in preclinical subjects or individuals with neurological diseases such as Probable Alzheimer's Disease (PRAD), Frontotemporal Dementias (FTD), Dementia with Lewy Bodies (DLB), Traumatic Brain Injury (TBI), and Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
The goal of this study is to examine olfactory function in preclinical subjects [n = 150] or individuals with neurological diseases such as Probable Alzheimer's Disease (PRAD) [n = 50], Mild Cognitive Impairment [n = 50], Frontotemporal Dementias (FTD) [n = 50], and Dementia with Lewy Bodies (DLB) [n = 50] that are part of the Longitudinal Research Cohort of the Massachusetts Alzheimer's Disease Research Center (IRB Protocol #: 1999P003693), are being treated by neurologists in the Memory Disorders or Movements Disorders Clinics at MGH, or are part of the community. The investigators will also examine individuals with Amyotrophic Lateral Sclerosis (ALS) [n = 50], ALS probands [n = 50], and ALS family controls [n = 50] that are part of the Neurological Clinical Research Institute (NCRI) protocols "NeuroBANK" (2013P001670), "Repository" (2006P000982), and "Longitudinal CSF" (2011P000785). Olfactory data will be correlated with existing data collected under the above-mentioned IRB protocols. The investigators will also be studying olfactory function in patients with mild TBI [n=50], and moderate and severe TBI [n=50], that are patients of Spaulding Rehabilitation Network. Specifically, the investigators will assess odor discrimination, odor identification, and episodic olfactory memory, using the OLFACT olfactometer run by a laptop or through a wireless iPad interface (Osmic Enterprises). Olfactory data collected from patients and age-matched control subjects [n = 100] will be correlated with existing structural MRI, functional MRI, and PET imaging data and with existing neuropsychological data collected under IRB protocols 1999P003693 and 2007P002107 ("Neurological Disease Registry"), NeuroBANK™ IRB protocol 2013P001670, Repository IRB protocol 2006P000982, and Longitudinal CSF IRB protocol 2011P000785.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Probable Alzheimer's Disease, prodromal Alzheimer's Disease, Frontotemporal Dementia, Mild Cognitive Impairment, or Dementia with Lewy Bodies or mild and moderate/severe TBI.
* Diagnosis of familial or sporadic ALS per El Escorial Criteria or individuals with known gene mutations associated with ALS (regardless of clinical phenotype).
* Age-matched controls
* Males and females with a minimum age of enrollment of 18 years. There is no maximum age of enrollment.

Exclusion Criteria:

* Primary pulmonary disease such as severe emphysema or asthma not under good medical control.
* Current sinusitis or common cold or upper respiratory infection, nasal polyps, or sinusitis.
* Traumatic or congenital anosmia
* Current or recent (past 6 months) alcohol or substance dependence. A prior history of alcohol or substance abuse will not be grounds for exclusion.
* Pregnancy
* Severe cognitive dysfunction
* Pneumocephalus
* Basilar skull fracture
* Known CSF leak
* Facial fractures to include Lefort I, II or III

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Diagnosis of Probable Alzheimer's Disease, prodromal Alzheimer's Disease, Frontotemporal Dementia, Mild Cognitive Impairment, or Dementia with Lewy Bodies or mild and moderate/severe TBI.
  2. Diagnosis of familial or sporadic ALS per El Escorial Criteria or individuals with known gene mutations associated with ALS (regardless of clinical phenotype).
  3. Age-matched controls
  4. Males and females with a minimum age of enrollment of 18 years. There is no maximum age of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-08-10 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Selective loss of episodic odor memory (Poor POEM status) will correlate with imaging and neuropsychological signs of neurodegenerative disease. | 9 years
  Poor POEM status determined by comparing the predicted POEM score with the actual POEM score will correlate with entorhinal cortical thickness, and neuropsychological test results.

SECONDARY OUTCOMES:
Correct responses on the episodic memory of odor percepts measure will correlate with entorhinal cortical thickness, and neuropsychological test results. | 9 years
  Compare number of trials correctly discriminated; compare number of odors correctly identified; and compare number of hits (accurate episodic memory of exposure to odor), and number of correct rejections (accurate episodic memory of non-exposure to odor). Correlate familiarity with number of hits and correct rejections.
Correct responses on the odor percept identification task will correlate with imaging and neuropsychological signs of neurodegenerative disease. | 9 years
  Compare number of trials of odors correctly identified will correlate with entorhinal cortical thickness, and neuropsychological test results.
Correct responses on the odor discrimination task will correlate with imaging and neuropsychological signs of neurodegenerative disease. | 9 years
  Compare number of trials correctly discriminated will correlate with entorhinal cortical thickness, and neuropsychological test results.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Albers, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dhilla Albers A, Asafu-Adjei J, Delaney MK, Kelly KE, Gomez-Isla T, Blacker D, Johnson KA, Sperling RA, Hyman BT, Betensky RA, Hastings L, Albers MW. Episodic memory of odors stratifies Alzheimer biomarkers in normal elderly. Ann Neurol. 2016 Dec;80(6):846-857. doi: 10.1002/ana.24792. Epub 2016 Nov 23. PMID 27696605